CLINICAL TRIAL: NCT05405764
Title: CONvalescence of FUntional Outcomes After ICU Stay by Oral Protein Supplementation
Brief Title: The CONFUCIUS Oral Protein Supplementation Trial
Acronym: CONFUCIUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion rate
Sponsor: ARH van Zanten (Other)
Collaborators: Intensive Care Research Foundation, Gelderse Vallei Hospital (Unknown); Rousselot BVBA (Industry)
Responsible Party: Sponsor-Investigator, ARH van Zanten, Prof. Dr. ARH van Zanten, MD, PhD, Gelderse Vallei Hospital
Organization: Gelderse Vallei Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL7915809121
Record Dates: First submitted 2022-04-13; First posted 2022-06-06 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Intensive Care Unit Acquired Weakness; Critical Illness
Keywords: Functional outcomes; Proteins; Intensive care unit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: parallel two-arm randomized blinded controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical non-transparent sachets with circle or square
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Porcine protein group (Experimental): The patients will receive protein supplements twice daily (2x22g) for a period of 6 weeks during breakfast and lunch. The supplement will be delivered in powdered form.
  Interventions: Dietary Supplement: Porcine protein supplement
- Carbohydrate group (Placebo Comparator): The patients will receive isocaloric carbohydrate supplements twice daily (2x21g) for a period of 6 weeks during morning and afternoon. The supplement will be delivered in powdered form.
  Interventions: Dietary Supplement: Control product maltodextrin supplement

INTERVENTIONS:
Dietary Supplement: Porcine protein supplement — Porcine protein supplementation
  Arms: Porcine protein group
Dietary Supplement: Control product maltodextrin supplement — Maltodextrin supplementation
  Arms: Carbohydrate group

SUMMARY:
Study the effect of 6-weeks porcine protein supplementation vs isocaloric comparator (carbohydrate) on functional outcomes in post ICU-patients. Patients will be included at ICU discharge. Included patients will receive the supplements twice daily (morning and afternoon), starting at the first day at the general ward.

To the best of our knowledge, a study on protein supplementation in the post-ICU period to address its effect on functional outcomes is lacking.

DETAILED DESCRIPTION:
Patients discharged from the Intensive Care Unit frequently suffer from Post Intensive Care Syndrome. This syndrome is characterized by muscle weakness and physical disabilities besides neurocognitive and psychological disturbances. Studies have shown that protein requirements in the post-ICU phase are often not met. Furthermore, protein supplementation in other patient groups have shown beneficial effects. However, a study on protein supplementation during the post-ICU period is lacking. This study aims to investigate the effect of protein supplementation on functional outcomes in post-ICU patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Living at home before hospital admission
3. Minimum ICU stay of 72 h
4. Informed consent

Exclusion Criteria:

1. MRC sum score ≤24 or 48≥ at ICU discharge
2. Barthel Index <14 before ICU admission
3. Chronic home ventilation
4. Mitochondrial or muscle disease or pareses
5. Serum creatinine > 173 mcmol/l (renal dysfunction)
6. Treatment limitations: DNR, no ICU readmission or palliative care
7. Inclusion in another intervention trial since ICU admission
8. Intolerance or allergy (for study products)
9. People living in a nursing home before hospital admission
10. Chronic Organizing Pneumonia or Pulmonary Interstitial Fibrosis
11. Inflammatory Bowel Disease
12. Diabetes Mellitus pharmaceutical medication at ICU admission
13. Underlying disease in which in the eyes of the attending physician, the protein or carbohydrate supplement could form a risk for the patient.
14. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Between group difference in composite score over time. The composite score consists of handgrip strength, muscle strength leg, muscle strength arm and exercise capacity. | At hospital discharge, an average of 11 days
  Between-group difference in physical function over time expressed as a composite score.
  The composite score consists of handgrip strength, muscle strength leg, muscle strength arm and exercise capacity.
  Handgrip strength will be measured with the Jamar dynamometer Muscle strength leg will be measured with the handheld dynamometer m. quadriceps fem.
  Muscle strength arm will be measured with the handheld dynamometer bicepss brachii Exercise capacity will be measured with the 6 minute walking distance test. Measured values will be compared to normative data. Calculated percentages will be added up and together form the composite score.
Between group difference in composite score over time. The composite score consists of handgrip strength, muscle strength leg, muscle strength arm and exercise capacity. | At the end of the intervention = 6 weeks after ICU discharge
  Between-group difference in physical function over time expressed as a composite score.
  The composite score consists of handgrip strength, muscle strength leg, muscle strength arm and exercise capacity.
  Handgrip strength will be measured with the Jamar dynamometer Muscle strength leg will be measured with the handheld dynamometer m. quadriceps fem.
  Muscle strength arm will be measured with the handheld dynamometer bicepss brachii Exercise capacity will be measured with the 6 minute walking distance test. Measured values will be compared to normative data. Calculated percentages will be added up and together form the composite score.
Between group difference in composite score over time. The composite score consists of handgrip strength, muscle strength leg, muscle strength arm and exercise capacity. | At 3-months follow-up
  Between-group difference in physical function over time expressed as a composite score.
  The composite score consists of handgrip strength, muscle strength leg, muscle strength arm and exercise capacity.
  Handgrip strength will be measured with the Jamar dynamometer Muscle strength leg will be measured with the handheld dynamometer m. quadriceps fem.
  Muscle strength arm will be measured with the handheld dynamometer bicepss brachii Exercise capacity will be measured with the 6 minute walking distance test. Measured values will be compared to normative data. Calculated percentages will be added up and together form the composite score.

SECONDARY OUTCOMES:
Handgrip strength | 6 weeks after ICU discharge (end of the intervention)
  Handgrip strength assessed with Jamar dynamometer
Muscle strength leg | 6 weeks after ICU discharge (end of the intervention)
  Muscle strength leg assessed with handheld dynamometer m. quadriceps fem.
Muscle strength arm | 6 weeks after ICU discharge (end of the intervention)
  Muscle strength arm assessed with handheld dynamometer m. biceps brachii
Exercise capacity | 6 weeks after ICU discharge (end of the intervention)
  Exercise capacity assessed with 6 minute walking distance
Lower extremity muscle strength | 6 weeks after ICU discharge (end of the intervention)
  Lower extremity muscle strength assessed with Timed chair stand test
Muscle strength and function (Chelsea Critical Care Physical Assessment Tool) | At hospital discharge, an average of 11 days
  CPAx is used to score physical morbidity. Score 0-50. The higher the score, the more independent.
Muscle strength and function (Medical Research Council-sumscore) | At hospital discharge (an average of 11 days), 6 weeks after ICU discharge (end intervention) and 3 months follow-up
  MRCsum is used to evaluate global muscle strength. Score from 0-60. The higher the score, the better the strength.
Functional performance | 6 weeks after ICU discharge (end intervention)
  Barthel score. Score 0-20. The higher the score, the more independent. Rockwood Clinical Frailty Scale. Score 1-9. The higher the score, the higher the frailty,
Health related quality of life | At hospital discharge (an average of 11 days), 6 weeks after ICU discharge (end intervention) and 3 months follow-up
  Health related quality of life assessed by EuroQol 5D
Muscle mass | At hospital discharge (an average of 11 days), 6 weeks after ICU discharge (end intervention) and 3 months follow-up
  Bio electric impedance analysis
Laboratory evaluation | 6 weeks after ICU discharge (end intervention)
  Plasma aminoacid concentrations
Clinical endpoint ICU readmission | 6 weeks after ICU discharge (end intervention) and 3 months follow-up
  Number of participants with ICU readmission after ICU discharge
Clinical endpoint hospital readmission | 6 weeks after ICU discharge (end intervention) and 3 months follow-up
  Number of participants with hospital readmission after hospital discharge
Clinical endpoint survival | 6 weeks after ICU discharge (end intervention) and 3 months follow-up
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Arthur RH van Zanten, MD, PhD, Principal Investigator — Gelderse Vallei Hospital
Locations (1):
- Gelderse Vallei Hospital, Ede, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paulus MC, Kouw IWK, Boelens YFN, Hermans AJH, Strookappe B, van Zanten ARH. Feasibility challenges in protein supplementation research: Insights from the convalescence of functional outcomes after intensive care unit stay in a Randomised Controlled Trial. Clin Nutr. 2025 Mar;46:119-130. doi: 10.1016/j.clnu.2025.01.020. Epub 2025 Jan 21. PMID 39914233
- [Derived] Boelens YF, Strookappe B, Vasse E, Mensink M, van Zanten AR. The effect of an intervention of porcine protein versus maltodextrin supplement on CONvalescence of FUnCtional outcomes after IcU Stay (CONFUCIUS): Study protocol for a randomized controlled, single-center, double-blind trial. Clin Nutr ESPEN. 2022 Dec;52:86-93. doi: 10.1016/j.clnesp.2022.10.008. Epub 2022 Oct 19. PMID 36513490